CLINICAL TRIAL: NCT00357942
Title: Local Administration of Morphine: An Evaluation of the Analgesic Effect at Stomatitis in Children
Brief Title: Topical Morphine for Stomatitis-related Pain Induced by Chemotherapy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Danish University of Pharmaceutical Sciences (Other)
Collaborators: Copenhagen University Hospital, Denmark (Other)
Responsible Party: Principal Investigator, Bettina Nygaard Nielsen, M.Sc. Pharm, sponsor contact person, Danish University of Pharmaceutical Sciences
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 102010; 2006-003260-53; 2006-003260-53 (EudraCT Number)
Record Dates: First submitted 2006-07-27; First posted 2006-07-28 (Estimated); Last update posted 2014-02-21 (Estimated); Status verified 2014-02

CONDITIONS: Pain; Mucositis
Keywords: Morphine; Mouthwash; Mucositis; Pain; Cancer; Child; Adolescent
MeSH Terms: conditions — Pain; Mucositis; Neoplasms | interventions — Injections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- C group I (Experimental): Morphine mouthwash and placebo i.v.(24 hours) Added on standard analgesic treatment (paracetamol and patient controlled analgesia, morphine)
  Interventions: Drug: morphine mouthwash; Drug: Placebo
- C group II (Active Comparator): Placebo mouthwash and morphine i.v.(24 hours) Added on standard analgesic treatment (paracetamol and patient controlled analgesia, morphine)
  Interventions: Drug: morphine solution for injection; Drug: Placebo
- C group III (Placebo Comparator): Placebo mouthwash and placebo i.v. (24 hours) Added on standard analgesic treatment (paracetamol and patient controlled analgesia, morphine)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: morphine solution for injection — morphine solution for injection 2 mg/ml, 50 microg/kg bodyweight, every 3 hour for 24 hours and placebo mouthwash
  Arms: C group II
Drug: Placebo — Placebo mouthwash
  Arms: C group II; C group III
Drug: morphine mouthwash — morphine mouthwash 2 mg/ml, 50 microg/kg bodyweight every 3 hour for 24 hours and placebo solution for injection
  Arms: C group I
Drug: Placebo — Placebo solution for injection every 3 hour for 24 hours
  Arms: C group I; C group III

SUMMARY:
Stomatitis/oral mucositis is a common side effect to chemotherapy. Stomatitis is often associated with painful ulcers in the mouth. The study hypothesis is that morphine administrated as a mouthwash can relieve stomatitis-related pain by a local analgesic effect.

The purpose of this study is to test the analgesic effect of a morphine mouthwash versus morphine injections or placebo (no active drug) in children/adolescents with stomatitis related to chemotherapy. Besides the investigational drugs (morphine mouthwash and morphine injections) the children/adolescents receive a standardized analgesic treatment for stomatitis-related pain.

ELIGIBILITY:
Inclusion Criteria:

* Children and adolescents at The Juliane Marie Center at Copenhagen University Hospital (Rigshospitalet, Denmark) or at The University Hospital in Lund (Sweden)
* Receiving chemotherapy in relation to a cancer disease
* Pain score of minimum 3 (VAS-scale) at rest for mouth pain in combination with stomatitis of minimum grade 1 (WHO-scale) or a pain score of minimum 5 (VAS-scale) at activity for mouth pain in combination with stomatitis of minimum grade 1 (WHO-scale)
* Negative pregnancy test, when relevant (judged by physician)
* Patients and/or parents understand and speak danish (Denmark) / swedish (Sweden)
* Signed informed consent

Exclusion Criteria:

* Allergic to the investigational medical product
* Alcohol or drug abuse

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2006-09; Primary Completion 2013-12 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Use of supplemental analgesics | 24 hours

SECONDARY OUTCOMES:
Pain score at rest | 24 hours
Pain score at activity (performance of oral hygiene) | 24 hours
Time to first dose of supplemental analgesics | 24 hours
Frequency and severity of side effects | 24 hours
Oral intake of food | 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Bettina N Nielsen, PhD student M.Sc.Pharm, Study Chair — Faculty of Pharmaceutical Sciences, University of Copenhagen
Locations (1):
- The Juliane Marie Center, Copenhagen University Hospital (Rigshospitalet), Copenhagen, Denmark